CLINICAL TRIAL: NCT00001689
Title: A Pharmacokinetic and Pharmacodynamic Study of Vincristine in Children With Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 980053; 98-C-0053
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-11

CONDITIONS: Acute Lymphocytic Leukemia; Leukemia
Keywords: Neurotoxicity; A.L.L.; Limited Sampling; Dose Individualization; Vinca Alkaloids
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Neurotoxicity Syndromes | interventions — Vincristine

INTERVENTIONS:
Drug: Vincristine

SUMMARY:
The pharmacokinetic behavior of vincristine in pediatric patients has not been well characterized. The present study will obtain detailed information on vincristine pharmacokinetics in patients being treated for standard risk ALL on CCG protocols 1952/1962. A limited sampling strategy will be developed, and the interpatient and intrapatient variability of vincristine pharmacokinetics in children will be studied. A correlation between vincristine neurotoxicity and vincristine pharmacokinetics will be sought.

DETAILED DESCRIPTION:
The pharmacokinetic behavior of vincristine in pediatric patients has not been well characterized. The present study will obtain detailed information on vincristine pharmacokinetics in patients being treated for standard risk ALL according to or on CCG protocols 1952/1962/1991. A limited sampling strategy will be developed, and the interpatient and intrapatient variability of vincristine pharmacokinetics in children will be studied. A correlation between vincristine neurotoxicity and vincristine pharmacokinetics will be sought.

ELIGIBILITY:
INCLUSION CRITERIA:

All patients 1 year and less than 10 years of age.

Patient must be diagnosed with acute lymphoblastic leukemia.

All CCG patients must be enrolled on CCG 1952, 1962 or 1991 protocols, or be treated according to a CCG standard risk ALL protocol. NCI patients must be treated according to CCG 1952 for the treatment of standard risk ALL. Enrollment onto the current trial (CCG B9802) should if possible take place concurrently with enrollment onto 1952/1962/1991 or start of treatment according to a CCG standard risk ALL protocol.

All patients or their legal guardians must sign a document of informed consent indicating their awareness of the investigational nature and the risks of this study.

EXCLUSION CRITERIA:

Previous underlying peripheral neuropathy.

Previous underlying central nervous system dysfunction.

Children with CNS toxicity attributable to other chemotherapeutic agents will not be followed with the Purdue pegboard test.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90
Dates: Start 1998-01; Study Completion 2003-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Crom WR, de Graaf SS, Synold T, Uges DR, Bloemhof H, Rivera G, Christensen ML, Mahmoud H, Evans WE. Pharmacokinetics of vincristine in children and adolescents with acute lymphocytic leukemia. J Pediatr. 1994 Oct;125(4):642-9. doi: 10.1016/s0022-3476(94)70027-3. PMID 7931891
- [Background] de Graaf SS, Bloemhof H, Vendrig DE, Uges DR. Vincristine disposition in children with acute lymphoblastic leukemia. Med Pediatr Oncol. 1995 Apr;24(4):235-40. doi: 10.1002/mpo.2950240405. PMID 7700168
- [Background] Adamson PC, Poplack DG, Balis FM. Pharmacology and drug resistance in childhood lymphoblastic leukemia. Hematol Oncol Clin North Am. 1990 Oct;4(5):871-94. PMID 2262483